CLINICAL TRIAL: NCT02648997
Title: An Open-Label Phase II Study of Nivolumab or Nivolumab/Ipilimumab in Adult Participants With Progressive/Recurrent Meningioma
Brief Title: An Open-Label Phase II Study of Nivolumab or Nivolumab/Ipilimumab in Adult Participants With Progessive/ Recurrent Meningioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, David Reardon, MD, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-490; CA209-324 (Other: BMS)
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Meningiomas
Keywords: Atypical Meningioma; Anaplastic Meningioma
MeSH Terms: conditions — Meningioma | interventions — Nivolumab; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Intervention Model Description: After completion of accrual to Cohort 1, we opened accrual to Cohort 2.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (original cohort): Nivolumab Monotherapy (Experimental): Nivolumab monotherapy (240 mg every 2 weeks)
  Interventions: Drug: Nivolumab - 240 mg
- Cohort 2 (Dose Level 0): Nivolumab in Combination with Ipilimumab (Experimental): * External Beam RT (IMRT, 3D-CRT, or proton-beam radiation therapy)
  * Followed by 4 cycles of Nivolumab (1 mg/kg every 3 weeks) + Ipilimumab (3 mg/kg every 3 weeks)
  * Followed by Nivolumab monotherapy (480 mg every 4 weeks).
  Interventions: Drug: Nivolumab - 240 mg; Drug: Nivolumab - 480 mg; Radiation: External Beam RT; Drug: Nivolumab - 1 mg/kg; Drug: Ipilimumab - 3 mg/kg
- Cohort 2 (Dose Level 0A): Nivolumab in Combination with Ipilimumab (Experimental): * External Beam RT (IMRT, 3D-CRT, or proton-beam radiation therapy)
  * Followed by 4 cycles of Nivolumab (3 mg/kg every 3 weeks) + Ipilimumab (1 mg/kg every 3 weeks)
  * Followed by Nivolumab monotherapy (480 mg every 4 weeks).
  Interventions: Drug: Nivolumab - 240 mg; Drug: Ipilimumab - 1 mg/kg; Drug: Nivolumab - 480 mg; Drug: Nivolumab - 3 mg/kg; Radiation: External Beam RT

INTERVENTIONS:
Drug: Nivolumab - 240 mg — 240 mg every 2 weeks
  Other Names: Opdivo; BMS-936558; ONO-4538
Drug: Ipilimumab - 1 mg/kg — 1 mg/kg every 3 weeks
  Other Names: BMS-734016; MDX010; MDX-CTLA4
  Arms: Cohort 2 (Dose Level 0A): Nivolumab in Combination with Ipilimumab
Drug: Nivolumab - 480 mg — 480 mg once every 4 weeks
  Other Names: Opdivo; BMS-936558; ONO-4538
  Arms: Cohort 2 (Dose Level 0): Nivolumab in Combination with Ipilimumab; Cohort 2 (Dose Level 0A): Nivolumab in Combination with Ipilimumab
Drug: Nivolumab - 3 mg/kg — 3 mg/kg every 3 weeks
  Other Names: Opdivo; BMS-936558; ONO-4538
  Arms: Cohort 2 (Dose Level 0A): Nivolumab in Combination with Ipilimumab
Radiation: External Beam RT — IMRT, 3D-CRT, or proton-beam radiation therapy
  Arms: Cohort 2 (Dose Level 0): Nivolumab in Combination with Ipilimumab; Cohort 2 (Dose Level 0A): Nivolumab in Combination with Ipilimumab
Drug: Nivolumab - 1 mg/kg — 1 mg/kg every 3 weeks
  Other Names: Opdivo; BMS-936558; ONO-4538
  Arms: Cohort 2 (Dose Level 0): Nivolumab in Combination with Ipilimumab
Drug: Ipilimumab - 3 mg/kg — 3 mg/kg every 3 weeks
  Other Names: BMS-734016; MDX010; MDX-CTLA4
  Arms: Cohort 2 (Dose Level 0): Nivolumab in Combination with Ipilimumab

SUMMARY:
This research study is studying targeted immunotherapies as a possible treatment for recurrent meningioma. The names of the study interventions involved in this study are nivolumab and ipilimumab.

DETAILED DESCRIPTION:
This research is a Phase II clinical trial, which means it will test the safety and effectiveness of nivolumab alone (Cohort 1) or in combination with ipilimumab (Cohort 2). Both nivolumab and ipilimumab are antibodies (types of human protein) that work to stop tumor cells from growing and multiplying by immunotherapy. Immunotherapy is trying to have the body's own immune system work against tumor cells.

Nivolumab and ipilimumab have both been used in other research studies and information from those other research studies suggests that these interventions may help to stop Meningioma cells from growing.

Nivolumab is FDA approved to treat other types of cancers, but the FDA (the U.S. Food and Drug Administration) has not yet approved this intervention for this type of cancer. The FDA has not approved the combination of nivolumab and ipilimumab for your specific disease, but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed WHO grade I, II or III meningioma that is progressive or recurrent. Metastatic meningiomas are allowed. Participants with grade I tumors must have failed radiation therapy.
* Prior therapy:
* There is no limit on the number of prior surgeries, radiation therapy, radiosurgery treatments or systemically administered therapeutic agents.

  * Patients may have been treated with standard external beam radiation or radiosurgery in any combination, however, an interval of ≥ 12 weeks (84 days) must have elapsed from the completion of the radiation therapy to start of study therapy unless there is histopathologic confirmation of recurrent tumor or there is new enhancing tumor outside the radiation field (beyond the high dose region or the 80% isodose line).
  * In addition, there must be subsequent evidence of tumor progression after completion of radiation therapy (grade I tumors only)
  * An interval of ≥ 28 days and full recovery (no ongoing safety issues) from surgical resection
  * An interval of ≥ 7 days from stereotactic biopsy;
* For prior systemic agents, participants must be at least 4 weeks (or 5 half-lives, whichever is shorter) from other prior cytotoxic chemotherapy (6 weeks from nitrosoureas) or biologic therapies.
* Participants must have recovered to grade ≤ 1 or pretreatment baseline from clinically significant adverse events related to prior therapy (exclusions include but are not limited to alopecia, laboratory values listed per inclusion criteria and lymphopenia);
* Be 18 years of age on day of signing informed consent.
* Have a Karnofsky performance status (KPS) ≥ 70 (Appendix A).
* Participants must demonstrate adequate organ and marrow function as defined below (all screening labs to be performed within 14 days of treatment initiation):

  * White blood cell (WBC) ≥ 2000/mm3
  * Absolute neutrophil count (ANC) ≥ 1,000/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 gm/dl
  * AST(SGOT)/ALT(SGPT) ≤ 3 x laboratory upper limit of normal (ULN)
  * Serum creatinine ≤ 1.5 X ULN OR
  * creatinine clearance (meas or calc) ≥ 60 mL/min for participants with creatinine levels > 1.5 X ULN
  * (GFR can be used in place of creatinine or creatinine clearance)
  * Total serum bilirubin ≤ 1.5 X ULN
  * (except participants with Gilbert's Syndrome, who can have a total bili < 5 X ULN)
  * Resting baseline oxygen saturation ≥ 92% at rest by pulse oximetry
* MRI (or CT if MRI contraindicated) within 14 days prior to start of study drug. Corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI or CT scan and the start of treatment, a new baseline MRI or CT is required.
* Ability to understand and the willingness to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study, including disease assessment by MRI (or CT), as confirmed by signing a written informed consent document.
* For cohort 2, patients must be a candidate for external beam radiotherapy including either conventional fractionated conformal dosing or stereotactic radiosurgical boost dosing (participants may enroll if they are receiving radiotherapy or have completed it within 8 weeks of starting immunotherapy);
* For cohort 2 patients who are undergoing fractionated conformal re-irradiation to a tumor site that has been previously irradiated, an interval of at least 6 months must have passed since they completed their prior irradiation to be eligible unless the current course of radiation is targeting a new area of tumor growth outside the 80% isodose line of the original radiation field as determined by the treating investigator.
* The effects of nivolumab on the developing human fetus are unknown. For this reason:
* Women of childbearing potential (WOCPB; defined in Section 3.4) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours of starting study therapy;
* Women must not be breastfeeding;
* WOCPB must agree to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study therapy plus 5 months after the last dose of Nivolumab.
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 7 months after the last dose of Nivolumab.
* Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly.
* At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:

  * HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

    * Male condoms with spermicide
    * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena by WOCBP subjects or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
    * Progestogen only hormonal contraception associated with inhibition of ovulation
    * Intrauterine hormone-releasing system (IUS)
    * Nonhormonal IUDs, such as ParaGard
    * Tubal ligation
    * Vasectomy
    * Complete Abstinence - Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.
  * LESS EFFECTIVE METHODS OF CONTRACEPTION

    * Diaphragm with spermicide
    * Cervical cap with spermicide
    * Vaginal sponge
    * Male Condom without spermicide
    * Progestin only pills by WOCBP subjects or male subject's WOCBP partner
    * Female Condom - A male and female condom must not be used together
  * UNACCEPTABLE METHODS OF CONTRACEPTION

    * Periodic abstinence (calendar, symptothermal, post-ovulation methods)
    * Withdrawal (coitus interruptus)
    * Spermicide only
    * Lactation amenorrhea method (LAM)
* NOTE: Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP participants must still undergo pregnancy testing as described.

Exclusion Criteria:

* Current or planned participation in a study of an investigational agent or using an investigational device.
* Tumors that are primarily localized to the brainstem or spinal cord;
* Evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan other than those that are grade ≤ 1 and either post-operative or stable on at least 2 consecutive MRI scans;
* Prior Therapy:
* Prior treatment with systemic immunosuppressive treatments, aside from systemic dexamethasone therapy for cerebral edema, such as methotrexate, chloroquine, azathioprine, etc. within 3 months of start of study therapy;
* Prior treatment with interstitial brachytherapy within 6 months of start of study therapy;
* All patients: Previous treatment with PD-1 or PD-L1 directed therapy;
* Cohort 2 patients: Previous treatment with CTLA-4 directed therapy;
* Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study;
* Minor surgical procedure (eg, stereotactic biopsy within 7 days of first study treatment; placement of a vascular access device within 2 days of first study treatment);
* Other Meds:
* Participants who are receiving any other investigational agents.
* Immunosuppressive medications / steroids:

  * Subject must not require high dose systemic corticosteroids defined as dexamethasone > 4 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks prior to Day 1of study therapy;
  * Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).
  * Physiologic replacement doses of systemic corticosteroids are permitted, even if > 10 mg/day prednisone equivalents.
  * A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Has received a live vaccine within 30 days prior to the first dose of study drug; seasonal influenza vaccination is permitted excluding the nasal spray formulation;
* No concurrent treatment on another clinical trial. Supportive care trials or non- treatment trials, e.g. quality of life, are allowed;
* Concomitant Medical Illnesses: Uncontrolled intercurrent illness, including-but not limited to:
* Known additional malignancy that is progressing or requires active treatment within 3 years of start of study drug. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy;
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis;
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results examples include but are not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements;
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition requiring hormone replacement, psoriasis not requiring systemic treatment, conditions not expected to recur in the absence of an external trigger or resolved childhood asthma/atopy would be exceptions to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study;
* Has an active infection requiring intravenous therapy;
* Positive test for hepatitis B virus surface antigen (HBV sAg) or detectable hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection
* Medical History:
* History of intracranial abscess within 6 months prior to start of study therapy;
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* NOTE: HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Nivolumab. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody;
* Prisoners or participants who are involuntarily incarcerated;
* Pregnant women are excluded from this study because Nivolumab is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Nivolumab, breastfeeding should be discontinued if the mother is treated Nivolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David A Reardon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Original Cohort): Nivolumab Monotherapy: Nivolumab monotherapy (240 mg flat dose) on Day 1 of every 2-week cycle
- Cohort 2 - Dose Level 0: Nivolumab in Combination With Ipilimumab: External Beam RT (IMRT, 3D-CRT, or proton-beam radiation therapy)
  Followed by 4 cycles of combination therapy: Nivolumab (1 mg/kg) + Ipilimumab (3 mg/kg) on Day 1 of every 3-week cycle
  Followed by Nivolumab monotherapy (480 mg flat dose) on Day 1 of every 4-week cycle
- Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab: External Beam RT (IMRT, 3D-CRT, or proton-beam radiation therapy)
  Followed by 4 cycles of combination therapy: Nivolumab (3 mg/kg) + Ipilimumab (1 mg/kg) on Day 1 of every 3-week cycle
  Followed by Nivolumab monotherapy (480 mg flat dose) on Day 1 of every 4-week cycle
Period: Overall Study
Arm/Group | Cohort 1 (Original Cohort): Nivolumab Monotherapy | Cohort 2 - Dose Level 0: Nivolumab in Combination With Ipilimumab | Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab
Started | 25 | 3 | 12
Completed | 25 | 3 | 11
Not Completed | 0 | 0 | 1
Not completed — Still receiving active study tx | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Original Cohort): Nivolumab Monotherapy | Cohort 2 - Dose Level 0: Nivolumab in Combination With Ipilimumab | Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab | Total
Number analyzed (Participants) | 25 | 3 | 12 | 40
Age, Customized [Count of Participants; unit: Participants]
  Age in years: 18-30 | 1 | 0 | 1 | 2
  Age in years: 31-40 | 2 | 0 | 1 | 3
  Age in years: 41-50 | 5 | 1 | 2 | 8
  Age in years: 51-60 | 6 | 1 | 3 | 10
  Age in years: 61-70 | 7 | 1 | 4 | 12
  Age in years: 71-80 | 2 | 0 | 1 | 3
  Age in years: 81-90 | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 1 | 5 | 20
  Male | 11 | 2 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 3 | 12 | 36
  Unknown or Not Reported | 4 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 23 | 3 | 10 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 3 | 12 | 40
Baseline Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — KPS Scale: 100 - Normal, no complaints, no evidence of dz; 90 - Able to carry on normal activity; minor signs/symptoms of dz; 80 - Normal activity w effort; some signs/symptoms of dz; 70 - Cares for self, unable to carry on normal activity/do active work; 60 - Requires occasional assistance, but able to care for most needs; 50 - Requires considerable assistance & frequent medical care; 40 - Disabled; requires special care & assistance; 30 - Severely disabled; hospitalization indicated; 20 - Very sick; hospitalization indicated; 10 - Moribund; fatal processes progressing rapidly; 0 - Dead.
  Participants
    70 | 8 | 1 | 2 | 11
    80 | 12 | 0 | 3 | 15
    90 | 5 | 2 | 5 | 12
    100 | 0 | 0 | 1 | 1
    UNK | 0 | 0 | 1 | 1
WHO Grade of Tumor at Registration [Count of Participants; unit: Participants] — The World Health Organization (WHO) classifies meningiomas into three main categories based on histopathologic findings including: grade I (benign); grade II (atypical); and grade III (anaplastic) meningiomas. Although most meningiomas are grade I and can be initially treated with surgery and/or radiation, effective therapy for those that recur or are either grade II (atypical) or grade III (anaplastic) remains elusive.
  Participants
    WHO Grade 2 | 18 | 2 | 7 | 27
    WHO Grade 3 | 7 | 1 | 4 | 12
    Unknown | 0 | 0 | 1 | 1
Current Recurrence # [Count of Participants; unit: Participants]
  1st Relapse | 1 | 1 | 6 | 8
  2nd Relapse | 12 | 2 | 3 | 17
  3rd Relapse | 4 | 0 | 0 | 4
  4th Relapse | 3 | 0 | 2 | 5
  Unknown | 0 | 0 | 1 | 1
  5th Relapse | 2 | 0 | 0 | 2
  6th Relapse | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Disease Progression At Six Months Following Initiation Of Study Therapy
Description: To evaluate the anti-tumor activity for single-agent nivolumab (cohort 1) or nivolumab plus ipilimumab following radiation therapy (cohort 2) among patients with recurrent/progressive grade I, II or III meningioma.
Time Frame: 6 months
Population: Subjects who withdrew consent to be followed or otherwise came off-study prior to reaching 6 months progression-free are not considered evaluable for PFS6 and are therefore not included here. This includes 2 COH 1 subjects and 1 COH 2 subject on Dose Level 0A. Another COH 2 subject on Dose Level 0A Withdrew consent to be followed without ever having received any study tx and is also not included in this dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Original Cohort): Nivolumab Monotherapy | Cohort 2 - Dose Level 0: Nivolumab in Combination With Ipilimumab | Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab
Number analyzed (Participants) | 23 | 3 | 10
Participants | 10 | 3 | 10

2. Secondary Outcome: Both Cohorts: Median Progression-Free Survival
Description: To evaluate additional measures of anti-tumor activity of single-agent nivolumab (cohort 1) and nivolumab plus ipilimumab after radiation therapy (cohort 2) among patients with recurrent/progressive grade I, II or III meningioma
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Both Cohorts: Median Overall Survival
Description: as for outcome 2
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Both Cohorts: Objective Radiologic Response Rate
Description: as for outcome 2
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Both Cohorts: Number of Participants With Treatment Related Adverse Events as Assessed by CTCAE v4.0.
Description: 1.2.1 To evaluate the safety and tolerability of single-agent nivolumab (cohort 1) and nivolumab plus ipilimumab after radiation therapy (cohort 2) among patients with recurrent/progressive grade I, II or III meningioma
Time Frame: 2 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Evaluate Circulating Immune Cell Subsets and Cytokines as Systemic Immune Correlative Markers
Description: Using fluorescence activated cell sorting (FACS), the absolute CD4 T cell count will be determined and phenotyping of T effector cells (CD4+CD69+) and T regulatory cells (CD4+CD25+FoxP3+) with determination of absolute number of naive, effector and regulatory T cells as well as percents/ratios of total population will also be determined. Soluble factors such as cytokines, chemokines, soluble receptors and antibodies to tumor antigens will be measured via commercially available multiplex assays and enzyme-linked immunosorbent assays (ELISA)
Time Frame: 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Evaluate Archival Tumor Expression of PD-L1 and PD-1 Expressing Tumor Infiltrating Lymphocytes
Description: To evaluate correlative biomarkers of systemic immune response among patients with recurrent/progressive grade II or III meningioma treated with single-agent nivolumab (cohort 1) and nivolumab plus ipilimumab after radiation therapy (cohort 2)
Time Frame: 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Evaluate Archival Tumor Expression of Immune Gene Expression Signature Utilizing the Nanostring Assay
Description: as for outcome 7
Time Frame: 2 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Assess Mean Changes From Baseline in the Level of Function Score for Each Domain of the Neurologic Assessment in Neuro-Oncology (NANO) Scale
Description: Evaluation Of Neurologic Function As Measured By The NANO Scale.
Time Frame: 2 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Determine Difference in Tumor Growth Rates Before and After Treatment That Would Allow Detection of Treatment Efficacy.
Description: Evaluation of change in tumor growth rate as measured by volumetric analysis
Time Frame: 2 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Determine if There Are Pre-treatment Predictors of Treatment Response Using Radiomic Analysis
Description: Evaluation of change in tumor growth rate as measured by volumetric analysis
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs are collected and reported from initiation of study medication through 30 days following the last dose of study medication. Any AE meeting Serious criteria (SAE) occurring anytime after a subject's consent through 100 days of the last dose of treatment are reported (or until the start of new anti-cancer treatment, whichever comes first) Adverse Events (AEs) monitored/assessed up to 4 years (as the maximum # of days a patient has been on active study treatment thusfar is 1258 days).
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered an investigational product; it does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product.
Groups:
- Cohort 1 (Original Cohort): Nivolumab Monotherapy: Nivolumab monotherapy (240 mg flat dose) on Day 1 of every 2-week cycle
  Note re: Reported # of Participants @ Risk:
  * Two COH 1 participants are not considered evaluable for 'All-Cause Mortality' because they withdrew consent to be followed.
  * One additional COH 1 participant is not considered evaluable for 'All-Cause Mortality' because they were lost to follow-up.
- Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab: External Beam RT (IMRT, 3D-CRT, or proton-beam radiation therapy)
  Followed by 4 cycles of combination therapy: Nivolumab (3 mg/kg) + Ipilimumab (1 mg/kg) on Day 1 of every 3-week cycle
  Followed by Nivolumab monotherapy (480 mg flat dose) on Day 1 of every 4-week cycle
  Notes re: Reported # of Participants @ Risk:
  * One COH 2 Dose Level 0A participant withdrew consent to be followed without ever having received any study tx and is therefore not included in the SAE, Other AE, or All-Cause Mortality datasets.
  * Two additional COH 2 Dose Level 0A participants are not considered evaluable for 'All-Cause Mortality' because they withdrew consent to be followed.
Arm/Group | Cohort 1 (Original Cohort): Nivolumab Monotherapy | Cohort 2 - Dose Level 0: Nivolumab in Combination With Ipilimumab | Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab
All-Cause Mortality (participants affected / at risk) | 20/22 | 2/3 | 1/9
Serious Adverse Events (participants affected / at risk) | 11/25 | 2/3 | 7/11
Other Adverse Events (participants affected / at risk) | 25/25 | 3/3 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Original Cohort): Nivolumab Monotherapy (N=25) | Cohort 2 - Dose Level 0: Nivolumab in Combination With Ipilimumab (N=3) | Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab (N=11)
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Adrenal Insufficiancy (Endocrine disorders) | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Endocrine disorders, other: Hypophysitis (Endocrine disorders) | 0 | 0 | 1
Endocrine disorders, other: Panhypopituitarism (Endocrine disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Death, NOS (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1
Fever (General disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
Infusion-related reaction (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other: Decline; PD (General disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Infections and infestations - Other: Bacteremia (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other: Pneumonia (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Cardiac troponin T increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 1
Edema cerebral (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Surgical and medical procedures - Other: Bone removal (Surgical and medical procedures) | 1 | 0 | 0
Surgical and medical procedures - Other: Craniotomy; Debulking Surgery (Surgical and medical procedures) | 3 | 0 | 0
Surgical and medical procedures - Other: Hardware removal (Surgical and medical procedures) | 1 | 0 | 0
Thromboembolic Event (Vascular disorders) | 0 | 0 | 2
Endocrine disorders - Other, specify: Panhypopituitarism (Endocrine disorders) | 0 | 1 | 0
Eye disorders - Other, specify: Left eye edema (Eye disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Original Cohort): Nivolumab Monotherapy (N=25) | Cohort 2 - Dose Level 0: Nivolumab in Combination With Ipilimumab (N=3) | Cohort 2 - Dose Level 0A: Nivolumab in Combination With Ipilimumab (N=11)
Anemia (Blood and lymphatic system disorders) | 5 | 0 | 3
Hypothyroidism (Endocrine disorders) | 2 | 2 | 2
Blurred vision (Eye disorders) | 4 | 0 | 1
Eye pain (Eye disorders) | 2 | 0 | 0
Eye disorders - Other, specify: Diplopia (Eye disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 6 | 0 | 5
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 1 | 5
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1
Fatigue (General disorders) | 16 | 3 | 8
Fever (General disorders) | 2 | 3 | 3
Sinusitis (Infections and infestations) | 3 | 0 | 0
Skin infection (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 0 | 0
Alanine aminotransferase increased (Investigations) | 9 | 2 | 6
Alkaline phosphatase increased (Investigations) | 4 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 1 | 5
Lipase increased (Investigations) | 6 | 1 | 3
Neutrophil count decreased (Investigations) | 5 | 1 | 2
Platelet count decreased (Investigations) | 3 | 1 | 1
Serum amylase increased (Investigations) | 8 | 0 | 2
White blood cell decreased (Investigations) | 3 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 2 | 7
Hypernatremia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 6 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 6 | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 3 | 0 | 0
Dysphasia (Nervous system disorders) | 2 | 0 | 2
Headache (Nervous system disorders) | 7 | 1 | 6
Paresthesia (Nervous system disorders) | 5 | 0 | 1
Seizure (Nervous system disorders) | 5 | 0 | 3
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Endocrine disorders - Other, specify: Testosterone deficiency (Endocrine disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Creatinine increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 4
Weight loss (Investigations) | 0 | 2 | 0
Investigations - Other, specify: Blood LDH increased (Investigations) | 0 | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1
Confusion (Psychiatric disorders) | 0 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders, Other; Specify: Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Endocrine disorders - Other, specify: TSH increased (Endocrine disorders) | 0 | 0 | 1
Eye disorders - Other, specify: Left field cut (Eye disorders) | 0 | 0 | 1
Eye disorders - Other, specify: Peripheral superior field cut (Eye disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 0 | 2
Facial pain (General disorders) | 0 | 0 | 1
Flu like symptoms (General disorders) | 0 | 0 | 3
Gait disturbance (General disorders) | 0 | 0 | 2
Infusion related reaction (General disorders) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other, specify: COVID + (Infections and infestations) | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Investigations - Other, specify: TSH increased (Investigations) | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders, Other: Specify - Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin/subcutaneous tissue disorders; Other, specify: Mild arm rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin/subcutaneous tissue disorders; Other, specify: Rash - fungal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02648997/Prot_SAP_000.pdf